CLINICAL TRIAL: NCT01831440
Title: The Influence of Pharmacotherapy and Psychotherapy for MDD After Remission on Psychology and Neuroimaging：A Comparative Longitudinal Study
Brief Title: Pharmacotherapy and Psychotherapy for MDD After Remission on Psychology and Neuroimaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ning Zhang, Vice-President of Nanjing Brain Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZKX10022
Record Dates: First submitted 2013-03-28; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Depressive Disorder
Keywords: depression; remission; Pharmacotherapy; psychotherapy; neuroimaging; psychology
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- medicine combined CBT (Other): Besides clinical routine antidepressant treatment,participants receive CBT weekly for 8 weeks and monthly until the end of the study.
  Interventions: Behavioral: medicine combined CBT
- medicine (SSRI antidepressants) (Other): clinical routine antidepressant treatment--Selective serotonin reuptake inhibitors（SSRIs）.
  Interventions: Drug: medicine

INTERVENTIONS:
Behavioral: medicine combined CBT — medicine：Clinical routine antidepressant treatment CBT：During the treatment period，weekly for 8 weeks，and monthly for the maintenance phase.Therapists receive group supervision monthly.
  Other Names: antidepressant combined cognitive-behavioral therapy
  Arms: medicine combined CBT
Drug: medicine — Participants receive only clinical routine antidepressant treatment,Which include fluoxetine (Prozac); sertraline (Zoloft); paroxetine (Paxil); citalopram (Celexa) ;escitalopram (Lexapro) and fluvoxamine (Luvox). It will be chosen according to special condition of every patient.
  Other Names: SSRI antidepressants
  Arms: medicine (SSRI antidepressants)

SUMMARY:
The purpose of this study is to determine the level of residual symptoms and psychosocial factors affecting recovery of psychosocial functions in MDD patients who reach remission, and investigate the recovery process of psychosocial functions.

The investigators suppose that even the patient is well-treated by drug,there are still many residual symptoms,and they also exist different degree of damage in the structure and functions of brain. CBT could help them obtain better recovery,especially in psychosocial functions.

DETAILED DESCRIPTION:
Objective:At present, clinical remission of depression is defined as a final HAMD score of less than 7. However, in clinical practice, the psychosocial functions of patients who reach remission are far from complete recovery. The recovery of psychosocial functions lags behind the disappearance of symptoms.so,we aim to determine the level of residual symptoms and psychosocial factors affecting recovery of psychosocial functions in MDD patients who reach remission, and investigate the recovery process of psychosocial functions.

Method:200 MDD patients who met the inclusion criteria were randomly divided into CBT group and control group.All of subjects would complete the psychological assessment at 0,1st,2nd,6th and 12th months for CBT group and 0,2nd,12th months for control group.ALL participants would undergo magnetic resonance imaging at 0,2nd,12th months.The scanning sequence is 3D,resting-state,task-state and diffusion tensor imaging（DTI）.During the magnetic resonance imaging（MRI） scans, subjects performed the facial and gender recognition tasks with three different facial stimuli(positive/neutral/negative).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of major depressive disorder (MDD)
* Hamilton Rating Scale for Depression(HAMD) less than 7

Exclusion Criteria:

* Bipolar disorder
* Substance dependence
* Neurological disorder or other mental disorder
* Severe body disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAMD） | one year
  The 24-item version of the Hamilton Rating Scale for Depression (HAMD; Hamilton, 1960) will be used for measuring severity of depressive symptoms.remission of depression is defined as a final HAMD score of less than 7.

SECONDARY OUTCOMES:
Magnetic Resonance Imaging | one year
  Scanning sequency：3D、resting-state、task-state、Diffusion Tensor Imaging（DTI） Task:explicit and implicit emotional processes.
The Beck Depression Inventory (BDI) | one year
  The Beck Depression Inventory (BDI), created by Dr. Aaron T. Beck, is a 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depression.
Generic Quality of Life Inventory-74 | one year
  Generic Quality of Life Inventory-74(GQOLI-74)created by Dr.Yang Desen and Dr. Li Lingjiang in 1998. It will be used for measuring the quality of life,efficacy and side effect.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Ning, Principal Investigator — Nanjing Brain Hospital
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Mattisson C, Bogren M, Horstmann V, Munk-Jorgensen P, Nettelbladt P. The long-term course of depressive disorders in the Lundby Study. Psychol Med. 2007 Jun;37(6):883-91. doi: 10.1017/S0033291707000074. Epub 2007 Feb 19. PMID 17306047
- [Background] Kuehner C. An evaluation of the 'Coping with Depression Course' for relapse prevention with unipolar depressed patients. Psychother Psychosom. 2005;74(4):254-9. doi: 10.1159/000085150. PMID 15947516
- [Background] Paykel ES, Scott J, Teasdale JD, Johnson AL, Garland A, Moore R, Jenaway A, Cornwall PL, Hayhurst H, Abbott R, Pope M. Prevention of relapse in residual depression by cognitive therapy: a controlled trial. Arch Gen Psychiatry. 1999 Sep;56(9):829-35. doi: 10.1001/archpsyc.56.9.829. PMID 12884889
- [Background] Watkins E, Scott J, Wingrove J, Rimes K, Bathurst N, Steiner H, Kennell-Webb S, Moulds M, Malliaris Y. Rumination-focused cognitive behaviour therapy for residual depression: a case series. Behav Res Ther. 2007 Sep;45(9):2144-54. doi: 10.1016/j.brat.2006.09.018. Epub 2007 Mar 26. PMID 17367751
- [Background] Petersen TJ. Enhancing the efficacy of antidepressants with psychotherapy. J Psychopharmacol. 2006 May;20(3 Suppl):19-28. doi: 10.1177/1359786806064314. PMID 16644768
- [Background] Vitiello B. Combined cognitive-behavioural therapy and pharmacotherapy for adolescent depression: Does it improve outcomes compared with monotherapy? CNS Drugs. 2009;23(4):271-80. doi: 10.2165/00023210-200923040-00001. PMID 19374457
- [Background] Scott J, Teasdale JD, Paykel ES, Johnson AL, Abbott R, Hayhurst H, Moore R, Garland A. Effects of cognitive therapy on psychological symptoms and social functioning in residual depression. Br J Psychiatry. 2000 Nov;177:440-6. doi: 10.1192/bjp.177.5.440. PMID 11059998
- [Derived] Zhong J, Xu J, Wang Z, Yang H, Li J, Yu H, Huang W, Wan C, Ma H, Zhang N. Changes in brain functional networks in remitted major depressive disorder: a six-month follow-up study. BMC Psychiatry. 2023 Aug 28;23(1):628. doi: 10.1186/s12888-023-05082-3. PMID 37641013
- See also: Click here for more information about Chinese Cognitive-Behavioral Therapy(CCBT) — http://www.cbtchina.com.cn/